CLINICAL TRIAL: NCT04956016
Title: Open-label Randomized Comparative Study of the Effects of a Classic High-frequency rTMS Treatment Versus a Deep rTMS Treatment in the Management of Resistant Depression
Brief Title: Effects of a Classic High-frequency rTMS Treatment Versus a Deep rTMS Treatment
Acronym: HAUVERDEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-A00796-35
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic rTMS treatment (Active Comparator): Arm A: classic rTMS treatment (use of the 8-shaped coil) and standard therapy
  Interventions: Device: classic rTMS using the 8-shaped coil
- treatment with deep rTMS (Active Comparator): Arm B: treatment with deep rTMS (use of the H1-shaped coil (helmet)) and standard therapies
  Interventions: Device: deep rTMS using the H1-shaped coil

INTERVENTIONS:
Device: classic rTMS using the 8-shaped coil — 20 rTMS sessions are planned (5 sessions per week)
  Arms: classic rTMS treatment
Device: deep rTMS using the H1-shaped coil — 20 rTMS sessions are planned (5 sessions per week)
  Arms: treatment with deep rTMS

SUMMARY:
The main objective is to demonstrate that dTMS is more efficient than high frequency rTMS with a conventional coil.

The patient will receive treatment arm A or B :

Arm A : classic rTMS treatment (use of the 8-shaped coil) and standard therapy Arm B: treatment with deep rTMS (use of the H-shaped coil (helmet)) and standard therapies.

20 rTMS sessions are planned (5 sessions per week) and 3 follow-up visits : at Day 30, Day 60 and Day 90.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects over 18 years old
* Having signed a free and informed consent
* Having a diagnostic of caracterised depressive episod recurrent or isolated according to DSM IV criteria (A.P.A 1994).
* Having an antidepressant treatment not modified since 3 weeks
* Score to MADRS scale ≥ 21
* Subject affiliated to a social security regimen

Exclusion Criteria:

* Depression with psychotic caracteristics
* Co-morbid diagnosis according to axis I (DSM IV) of schizophrenia, dependence (or abuse) on alcohol and / or another substance (lifetime)
* Patient who has already undergone seismotherapy for current episode and non-responder to this treatment
* Patient hospitalized under duress or under legal protection (guardianship, curatorship)
* Patient with a high risk of suicide (item 10 of MADRS > 4) in the absence of hospitalization.
* Contra-indication for IRM exam or rTMS : personnal history of comitial crisis, of neurological or neurochirurgical pathologies, metallic prosthetic material or foreign body (pacemaker, intraoculare ferromagnetic material, implanted cardiac defibrillator, cochlear implant, metal clip
* Pregnancy
* Simultaneous participation to another interventionnal study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
A 50% change of MADRS score | Day 60
  The main objective is to demonstrate that dTMS is more efficient than high frequency rTMS with a conventional coil.
  Modification of the MADRS score compared to baseline score. MADRS stands for Montgomery-Asberg Depression Rating Scale. It is used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. A score from 0 to 6 being normal/symptom absent and a score >34 being severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ghina HARIKA-GERMANEAU, Dr, Principal Investigator — Centre Hospitalier Henri Laborit
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France